CLINICAL TRIAL: NCT06003296
Title: Calcaneocuboid Arthrodesis in Triple Arthrodesis by Plate Versus Screw: Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrazik Talaat Abdelrazik Khalifa, Assiut, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Calcaneocuboid arthrodesis
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Calcaneocuboid Osteoarthritis Secondary to Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screw fixation (Other): Calcaneocuboid arthrodesis in triple arthrodesis by Screw fixation
  Interventions: Procedure: Calcaneocuboid arthrodesis

INTERVENTIONS:
Procedure: Calcaneocuboid arthrodesis — Calcaneocuboid arthrodesis in triple arthrodesis

SUMMARY:
Investigators aim to compare clinical and radiological outcome of use of plate versus screw fixation for calcaneocuboid arthrodesis in adult population.

DETAILED DESCRIPTION:
The calcaneocuboid joint is stable, even although multiple conditions might affect the joint, ranging from osteoarthritis to fracture, subluxation, and dislocation. Calcaneocuboid arthrodesis is more commonly performed as an adjunct procedure with other rearfoot procedures such as triple arthrodesis and is less used as isolated fusion.[1],[2],[3] What the most effective and least cost method for calcaneocuboid arthrodesis?! Many conditions that may affect foot that cause pain ; and there are many methods for relieve that pain , one of these is arthrodesis , and calcaneocuboid joint one of the most affected joints , and commonly we do calcaneocuboid arthrodesis as a part of triple arthrodesis ( subtalar , talonavicular , calcaneocuboid ); The traditional fixation for a calcaneocuboid (CC) arthrodesis in triple arthrodesis is with a 6.5-mm cancellous screw. This procedure can be technically challenging. Fixation with a locking compression plate (LCP) may be easier to perform while achieving compression perpendicular to the fusion site. Investigators suppose that plate is more powerful than screw in calcaneocuboid arthrodesis. The purpose of this study was to compare the load to failure and the stiffness for each fixation method. [4],[5],[6] literature reveal that: More stability to the fusion site can be applied by using plate fixation. Rationale of the research that: calcaneocuboid arthrodesis with screw is effective and least cost compare to plate fixation? [7]

ELIGIBILITY:
Inclusion Criteria:

all patients who will be operated by calcaneocuboid fusion for any indication age range 18-65 no paralytic patients

Exclusion Criteria:

* age < 18 , > 65 acute calcaneal fracture infection non union bone defect that need bone graft refusing to participate in the study neuropathic patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Assess calcaneocuboid arthrodesis union | One year
  calcaneocuboid arthrodesis union by RUST score

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrazik Talaat, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt